CLINICAL TRIAL: NCT06817421
Title: Immunogenicity of Opportunistic Pneumococcal Conjugate Vaccination (Pneumosil®) Versus Control (Typhoid Conjugate Vaccine, Typbar TCV®) in Children Aged 6-59 Months Hospitalised With Severe Acute Malnutrition: a Single-centre, Double-blind, Randomised Controlled Trial in Timor-Leste
Brief Title: Opportunistic Pneumococcal Immunisation Trial in MALnutrition
Acronym: OPTIMAL
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nick Fancourt (Other)
Collaborators: Murdoch Childrens Research Institute (Other); The University of Western Australia (Other); University of Edinburgh (Other); Timor-Leste Ministry of Health (Unknown)
Responsible Party: Sponsor-Investigator, Nick Fancourt, Senior Research Fellow, Menzies School of Health Research
Organization: Menzies School of Health Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MENTL2024-4996; U1111-1312-6848 (Other: WHO)
Record Dates: First submitted 2025-01-28; First posted 2025-02-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Severe Acute Malnutrition in Childhood; Pneumococcal Disease; Pneumococcal Vaccines; Pneumococcal Infection; Pneumonia in Children
Keywords: Pneumococcal; Severe Acute Malnutrition in childhood; Pneumococcal vaccine; Pneumosil; Pneumococcal disease; Pneumococcal infection; Pneumonia
MeSH Terms: conditions — Pneumococcal Infections; Pneumonia | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Intervention Model Description: A prospective, single-centre, double-blind, phase 4, randomised, controlled trial in children aged 6-59 months hospitalised with severe acute malnutrition.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm: Pneumosil (Experimental)
  Interventions: Biological: Pneumococcal conjugate vaccine
- Control Arm: Typbar TCV (Other)
  Interventions: Biological: Typhoid conjugate vaccine

INTERVENTIONS:
Biological: Pneumococcal conjugate vaccine — 10-valent pneumococcal polysaccharide conjugate vaccine at a dosage of 2μg for each serotype polysaccharide for 1, 5, 6A, 7F, 9V, 14, 19A, 19F, 23F, and 4μg for serotype 6B, conjugated to a carrier protein (CRM197), polysorbate 20 and aluminium phosphate as an adjuvant. Administered as an intramuscular injection of 0.5mL.
  Arms: Treatment Arm: Pneumosil
Biological: Typhoid conjugate vaccine — Typhoid conjugate vaccine at a dosage of 25μg purified Vi capsular polysaccharide of Salmonella typhi Ty2 conjugated to Tetanus Toxoid with preservative (2-Phenoxyethanol). Administered as an intramuscular injection of 0.5mL.
  Arms: Control Arm: Typbar TCV

SUMMARY:
The goal of the OPTIMAL clinical trial is to learn if a dose of a pneumococcal conjugate vaccine (PCV) generates a good immune response in young children who are in hospital with severe acute malnutrition.

Researchers will compare an intervention group who get a dose of a PCV (Pneumosil) to a control group who get a dose of a Typhoid conjugate vaccine (Typbar TCV). To ensure all participants receive timely potential benefits, at 3 months participants in the intervention group with receive a dose of Typbar TCV, and those in the conrol group will receive a dose of Pneumosil.

Participants will be visited 4 times at their homes over six months after vaccination, with a phone review at 12 months after vaccination.

DETAILED DESCRIPTION:
This is a prospective, single-centre, double-blind, randomised controlled trial in 264 children aged 6-59 months hospitalised with severe acute malnutrition.

Participants will be randomised (1:1) to receive either a dose of a pneumococcal conjugate vaccine (Pneumosil, the intervention group) or a dose of a Typhoid conjugate vaccine (Typbar TCV, the control group). Stratification for randomisation will be done on (a) prior immunisation with a PCV (confirmed or unknown/unvaccinated); and (b) severity of malnurition (weight-for-height/length z-score <-4 or >=-4). Participants will be enrolled as soon as practical after admission to hospital, while randomisation and vaccine administration will occur once the participant is medically stable in the 'transition phase' of SAM care.

The primary objective is to demonstrate that immune responses to the 10 pneumococcal serotypes in Pneumosil are better in participants who receive Pneumosil, compared to those who receive Typbar TCV, when measured 28 days after vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 6-59 months at the time of hospitalisation
2. Hospitalised with severe acute malnutrition (SAM, defined as any one of a, b, or c):

   1. weight-for-length/height z-score <-3; or
   2. middle upper arm circumference <11.5cm; or
   3. bilateral pitting pedal oedema unexplained by other causes
3. Parent/carer is willing for their child to participate in the study and has provided written informed consent
4. Parent/carer is willing to comply with all study procedures outlined in the protocol, including specimen collection, for the duration of the study

Exclusion Criteria:

1. Known history of allergy or hypersensitivity to any component of either study vaccine, including diphtheria toxoid, or a history of anaphylactic shock.
2. Treatment with another investigational drug or other intervention in the 30 days prior to randomisation, or ongoing participation in another clinical trial.
3. Suspected primary or secondary immunodeficiency or prolonged administration (>14 days) of an immune modifying drug (including oral glucocorticoids) in the past 3 months.
4. Known terminal illness expected to result in death within 6 months.
5. Participants who, in the opinion of the site Principal Investigator, are unable to comply with the study protocol, including scheduled visits, assessments, and any other protocol-required procedures.
6. Previously enrolled in this trial.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 214 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Serotype-specific immunoglobulin G (IgG) antibodies | 4 weeks after vaccination
  Pneumosil serotype-specific (1, 5, 6A, 6B, 7F, 9V, 14, 19A, 19F, 23F) immunoglobulin G (IgG) geometric mean concentrations (GMCs).

SECONDARY OUTCOMES:
Serotype-specific IgG antibodies | 4 weeks and 3 months after vaccination
  Pneumosil serotype-specific IgG GMCs
Proportion of participants with serotype-specific IgG antibody responses ≥ 0.35 μg/mL | 4 weeks and 3 months after vaccination
  Proportion of participants with Pneumosil serotype-specific IgG concentrations ≥ 0.35μg/mL
Functional antibody responses | 4 weeks and 3 months after vaccination
  Pneumosil serotype-specific pneumococcal geometric mean opsonisation indices (GMOIs)
Functional antibody responses | 4 weeks and 3 months after vaccination
  Proportion of participants with Pneumosil serotye-specfiic pneumococcal opsonisation indices (OIs) >8
Salivary IgG antibodies | 4 weeks and 3 months after vaccination
  Serotype-specific salivary IgG (μg/ml) for Pneumosil serotypes and non-vaccine types 3, 4, 11A, and 18C
Salivary immunoglobulin A (IgA) antibodies | 4 weeks and 3 months after vaccination
  Serotype-specific salivary IgA (μg/ml) for Pneumosil serotypes and non-vaccine types 3, 4, 11A, and 18C
Nasopharyngeal carriage of pneumococcus | 3 months after vaccination
  Proportion of participants with nasopharyngeal carriage of Pneumosil vaccine-type pneumococci and their antimicrobial resistance patterns
Severe acute malnutrition recovery | Reviewed at all study visits until completion (12 months after vaccination)
  Weight-for-height/length z-score >= -2 or MUAC >12.5cm
Re-hospitalisation | 3 months and 12 months after vaccination
  Any repeat admission to hospital as confirmed by medical records
Mortality | 3 and 12 months after vaccination
  Deaths as reported. Cause of death determined from review of medial records.
Composite illness or mortality | Reviewed at all study visits until completion (12 months after vaccination)
  Repeat hospitalisation(s) or death.
Salmonella Typhi antibodies | 4 weeks and 3 months after vaccination for all participants, plus 4 months and 6 months after vaccination for participants in the control arm
  Proportion of paticipants with >4 fold rise (compared to pre-vaccination) of Salmonella Typhi anti-Vi IgG geometric mean titres (GMTs)

CONTACTS AND LOCATIONS:
Locations (1):
- Guido Valadares National Hospital (HNGV), Dili, Timor-Leste, Timor-Leste

IPD SHARING:
Plan to Share IPD: Undecided
Plan for IPD sharing is in development.

REFERENCES:
- See also: Pneumosil product information — https://extranet.who.int/prequal/vaccines/p/pneumosilr-0
- See also: Typbar-TCV product information — https://extranet.who.int/prequal/vaccines/p/typbar-tcv-0